CLINICAL TRIAL: NCT03496805
Title: A Phase 2 Double-blind, Placebo-controlled Study of the Effects of Muscadine Grape Extract in Men With Prostate Cancer on Androgen Deprivation Therapy
Brief Title: Effects of Muscadine Grape Extract in Men With Prostate Cancer on Androgen Deprivation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00047840; CCCWFU 85417 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Prostate Cancer
Keywords: Muscadine Grape Extract; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study. Only the lead-site investigational pharmacy team and the statistician will unblinded. The blind will be maintained until the study is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MGE group (Experimental): Patients will be randomized to muscadine grape extract (MGE). The patients will take 4 capsules by mouth BID (twice daily). Androgen deprivation therapy (ADT) is to be started within 60 days prior to initiation of MGE.
  Interventions: Drug: MGE; Other: ADT
- Placebo group (Placebo Comparator): Patients will be randomized to placebo. The patients will take 4 capsules by mouth BID (twice daily). Androgen deprivation therapy (ADT) is to be started within 60 days prior to initiation of placebo.
  Interventions: Other: Placebo; Other: ADT

INTERVENTIONS:
Drug: MGE — The patients will take 4 capsules by mouth BID (twice daily).
  Arms: MGE group
Other: Placebo — The patients will take 4 capsules by mouth BID (twice daily).
  Arms: Placebo group
Other: ADT — Androgen deprivation therapy (ADT) is to be started within 60 days prior to initiation of MGE.

SUMMARY:
It is estimated that one-third of the more than 7 million deaths from cancer worldwide are attributable to potentially modifiable risk factors, with 374,000 deaths preventable through diet modification alone. Diet supplementation for the prevention or treatment of cancer is attractive, as implementation is relatively easy, even in populations with reduced incomes and resources. Grape extracts or active components isolated from grapes have received attention as chemopreventive or therapeutic agents based upon their anti-proliferative, anti-inflammatory, and anti-oxidant properties. Evidence from preclinical trials also suggests that muscadine grape products may decrease systemic inflammation. This study builds upon promising preclinical and clinical evidence to determine if the addition muscadine grape extract (MGE) to androgen deprivation therapy (ADT) improves symptoms in men with prostate cancer.

DETAILED DESCRIPTION:
Primary Objective: To compare levels of fatigue in the MGE group compared to the placebo group at 6 months.

Secondary Objectives

* To compare levels of fatigue in the MGE group compared to the placebo group at 3, 9, and 12 months.
* To compare quality of life in men in the MGE group compared to the placebo group.
* To compare physical function, physical fitness, and body composition in men in the MGE group compared to the placebo group.
* To compare time to PSA progression (from study entry) in men in the MGE group compared to the placebo group.
* To compare progression-free survival (from study entry) in men in the MGE group compared to the placebo group.

OUTLINE: Participants are randomized into 1 of 2 groups.

GROUP I (Muscadine grape extract): Participants begin Androgen deprivation therapy prior to receiving muscadine grape extract and then receive muscadine grape extract orally (PO) twice daily (BID) for 12 months in the absence of disease progression or unacceptable toxicity.

GROUP II (PLACEBO): Participants begin Androgen deprivation therapy prior to receiving placebo and then receive placebo PO BID for 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 72 hours and then for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Men age ≥18 years who are fluent in English.
* Histologically confirmed prostate adenocarcinoma.
* Prior surgical castration or active ongoing use of androgen deprivation therapy (ADT) with expectation by the treating physician that patient would remain on ADT for the upcoming 12 months. ADT in the setting of definitive radiation therapy permitted. Concurrent treatment with androgen pathway inhibitors (examples include enzalutamide, abiraterone, darolutamide, apalutamide) permitted..
* Normal organ and marrow function function (labs within 30 days prior to study entry) as defined below:

White blood cell count greater than or equal to 3,500/mcL (or 3.5 (x103)) Platelet count greater than or equal to 75,000/mcL (or 75 (x103)) Hemoglobin greater than or equal to >9 g/dL Total bilirubin less than or equal to 2.5 X institutional upper limit of normal AST(SGOT)/ALT(SGPT) less than or equal to 2.5 X institutional upper limit of normal Creatinine less than or equal to 2.5 X institutional upper limit of normal

* Able to ambulate (use of assist device is acceptable).
* Able to cooperate with study-related activities.
* The effects of MGE on the developing human fetus are unknown. Men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Symptomatic metastatic disease requiring medical treatment (i.e., painful metastases to bone).
* Prostate cancer related surgery or radiation within 60 days prior to study entry.
* Documented rise in PSA (defined as rise of > 0.5 ng/mL) while on current prostate cancer therapy, determined by PSA values, at least one of which must be during the 6 months prior to study entry PSA values must be at least 7 days apart.
* Planned cessation of ADT or planned use of cytotoxic chemotherapy (i.e., docetaxel) within 12 months after study entry.
* Ongoing use of any other investigational cancer-directed agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MGE.
* Inability to swallow oral medications.
* Malabsorption due to bowel resection or gastrointestinal disease leading to uncontrolled diarrhea, or persistent nausea or vomiting requiring daily antiemetic therapy for symptom management within the past week.
* Uncontrolled intercurrent illness, including but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Changes in fatigue | Baseline and 6 months
  The PROMIS Fatigue 7a Short-Form assesses the experience (3 items) and impact (4 items) of fatigue. Item responses are rated on a five-point scale ranging from "never" to "always" and are summed for a total score and transformed to a T-score metric. Higher scores indicate more fatigue. Recommendations for classifying fatigue based on the T scores are as follows: <50 normal; 50-59 mild; 60-69 moderate; ≥70 severe.

SECONDARY OUTCOMES:
Changes in quality of life: PROMIS | Baseline and 6 months
  General Quality of Life will be measured using the Patient Reported Outcomes Measurement Information System© (PROMIS©) Global Health Short Form (SF), a 10-item instrument representing multiple domains. Items assess self-reported measures of general aspects of physical, mental and social health in adults. Raw scores are summed within each sub-domain, and converted to T-scores. Higher scores indicate better general health than the general population.
Changes in quality of life: HFRDIS | Baseline and 6 months
  Quality of life will be assessed by the Hot Flash Related Daily Interference Scale (HFRDIS). HFRDIS is a 10-item scale that assesses the degree to which hot flashes interfere with a variety of daily activities and quality of life. Interference is rated on an 11-point scale (0=not interfere; 10=completely interfere). Higher scores indicate more interference.
Changes in sleep disturbance | Baseline and 6 months
  Sleep disturbance will be measured using the PROMIS Sleep Disturbance (SD) SF 8a. The PROMIS-SD items assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. Each question has five response options ranging in value from one to five. The lowest possible raw score is 8; the highest possible raw score is 40. Raw scores are converted to a standardized T-score. Higher scores indicate more sleep disturbance.
Changes in cognitive abilities | Baseline and 6 months
  Cognitive abilities will be measured using the PROMIS Cognitive Abilities SF 4a, which assesses patient-perceived functional abilities related to mental acuity, concentration, and memory. Raw scores are converted to a standardized T-score; final scores are represented by the T-score. Higher scored indicate more cognitive ability.
Changes in self-reported physical function | Baseline and 6 months
  Self-reported physical function will be measured using the PROMIS Physical Function 10a SF, which is designed to assess self-reported capability rather than actual performance of physical activities. The form consists of 10 items. Raw scores are summed within each sub-domain, and converted to T-scores. Higher scores indicate better physical function general health than the general population.
Changes in physical performance | Baseline and 6 months
  Physical performance will be objectively assessed using the Short Physical Performance Battery (SPPB). Each performance measure is scored ranging from 0-4 (0 = unable to complete; 4 = highest performance level), with total sum score range from 0-12. Lower score on the SPPB have been associated with increased risk of disability, hospitalization and worse survival among older adults with and without cancer.
Changes in sub-maximal exercise | baseline and 6 month
  Submaximal (6-minute walk) exercise capacity will be measured to assess physical fitness.
Changes in body composition | Baseline and 6 months
  Whole body lean mass, fat mass, and bone mass will be measured by duel energy X-ray absorptiometry (DXA). BMI will be calculated from height and weight.
Changes in prostate-specific antigen (PSA) progression | baseline, 6, and 12 months
  PSA will be measured at baseline, 6, and 12 months while patient is on MGE/placebo.
Progression-free survival | up to 12 months
  Progression-free survival is defined as the time from initiation of ADT treatment to disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Klepin, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - WG Hefner VA Medical Center, Salisbury, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT03496805/ICF_000.pdf